CLINICAL TRIAL: NCT03111368
Title: Endoscopic Ultrasound-guided Fine Needle Aspiration (EUS-FNA) of Solid Pancreatic Mass: Comparison Between Negative Pressure and Slow-pull Technique
Brief Title: EUS-FNA of Solid Pancreatic Mass: Comparison Between Negative Pressure and Slow-pull Technique
Acronym: EUS-FNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry); Medi - Globe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 41620315.9.0000.0068
Record Dates: First submitted 2016-04-01; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2016-06

CONDITIONS: Pancreatic Neoplasm
Keywords: eus-fna; pancreatic neoplasm; slow-pull; negative pressure
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EUS- FNA Slow-pull (Active Comparator): Endoscopic ultrasound-guided fine needle aspiration using a stylet slow-pull technique of solid pancreatic mass
  Interventions: Procedure: Endoscopic ultrasound-guided fine needle aspiration
- EUS-FNA Negative Pressure (Active Comparator): Endoscopic ultrasound-guided fine needle aspiration using negative pressure technique of solid pancreatic mass
  Interventions: Procedure: Endoscopic ultrasound-guided fine needle aspiration

INTERVENTIONS:
Procedure: Endoscopic ultrasound-guided fine needle aspiration — pancreatic solid mass punctured with a 22G endoscopic ultrasound needle
  Other Names: EUS-FNA

SUMMARY:
50 patients with pancreatic mass will undergo endoscopic ultrasound-guided fine needle aspiration using two techniques: negative pressure and slow-pull. Cytological results will be compared.

DETAILED DESCRIPTION:
The study will analyze the cytological results of endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) of pancreatic mass using two different techniques of needle suction. Negative pressure and slow-pull. 50 patients with pancreatic mass will be submitted to four passes with both techniques. Each patient will be randomized to decide which technique will be first and subsequently on a alternated fashion until four passes are completed. Smear cytology and cell block preparations for each technique were obtained. The pathologist was blinded for the EUS-FNA technique.

ELIGIBILITY:
Inclusion Criteria:

* pancreatic solid mass

Exclusion Criteria:

* endoscopic ultrasound non accessible lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2016-06-23 (Actual); Study Completion 2016-06-23 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | 24 months
  cytological results after endoscopic ultrasound fine needle aspiration

CONTACTS AND LOCATIONS:
Overall Officials: Spencer Cheng, Principal Investigator — Hospital das Clinicas Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Hospital das Clinicas da FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No